CLINICAL TRIAL: NCT06604806
Title: Comparison of Postoperative Analgesic Efficacy of Quadroiliac Plane Block and Pericapsular Nerve Group (PENG) Block in Femoral Fractures: A Multicenter Randomized Controlled Prospective Study
Brief Title: Comparison of Quadroiliac Plane Block and Pericapsular Nerve Group (PENG) Block in Femoral Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Engin Ihsan Turan, M.D., Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: QIP-PFN
Record Dates: First submitted 2024-09-17; First posted 2024-09-20 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Femur Fractures
Keywords: postoperative pain management; fascial plan blocks; pain; analgesia
MeSH Terms: conditions — Femoral Fractures; Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- opioid consumption (Active Comparator): opioid consumption of the patients in patient controlled analgesia device
  Interventions: Procedure: PENG Block; Procedure: Quadro-Iliac plane block
- Visual Analogue Scale scores of the patients (Active Comparator): Visual Analogue Scale scores of the patients
  Interventions: Procedure: PENG Block; Procedure: Quadro-Iliac plane block

INTERVENTIONS:
Procedure: PENG Block — With the patient in the supine position, the ultrasound probe is placed transversely over the anterior superior iliac spine (ASIS). After identifying the ASIS, the transducer is aligned with the pubic ramus and rotated approximately 45 degrees to become parallel to the inguinal crease. The transducer is moved medially until the anterior inferior iliac spine (AIIS), iliopubic eminence (IPE), and psoas tendon are clearly visualized as anatomical landmarks. After confirming the correct location with saline injection, 50 mg of 0.25% bupivacaine will be administered.
Procedure: Quadro-Iliac plane block — With the patient in the prone position, a low-frequency convex transducer (2-6 MHz) and a 22G x 100 mm peripheral nerve block needle (Stimuplex® Ultra 360®, B-Braun) will be used. The transducer will be placed transversely at the L3 level to identify the spinal processes, followed by lateral movement to visualize the transverse process within the erector spinae muscle. The transducer will then be rotated parasagittally and moved caudally to locate where the Quadratus Lumborum muscle (QLM) attaches to the iliac crest. After confirming the location with saline, 50 mg of 0.25% bupivacaine will be administered under the fascia of the QLM.

SUMMARY:
This prospective, multicenter study will compare the postoperative analgesic efficacy of the Quadroiliac Plane Block (QIPB) and Pericapsular Nerve Group (PENG) block in patients undergoing femoral neck fracture surgery. Eligible patients will be randomly assigned to receive one of the blocks postoperatively under spinal anesthesia. The blocks will be administered by experienced anesthesiologists, and informed consent will be obtained from all participants.

Pain levels will be assessed using the visual analog scale (VAS) at rest and during movement at 0, 6, 12, and 24 hours post-surgery. Opioid consumption will be recorded through patient-controlled analgesia (PCA), and any need for rescue analgesia will be evaluated. Routine postoperative pain management will also include intravenous paracetamol.

DETAILED DESCRIPTION:
This prospective, multicenter, observational study will be conducted at Başakşehir Çam and Sakura City Hospital and Kanuni Sultan Süleyman Training and Research Hospital. The study will include patients aged 18 and older, with an ASA score of I-II-III, undergoing femoral neck fracture surgery under spinal anesthesia. Patients with no history of bleeding diathesis, anticoagulant use, or allergies to the drugs used in the study, and without neuropathic diseases such as diabetes mellitus, will be randomly assigned to receive either the Pericapsular Nerve Group (PENG) block or the Quadroiliac Plane Block (QIPB) postoperatively.

Informed consent will be obtained from all patients, and detailed explanations of both blocks will be provided. Randomization will be performed using a computer program, assigning patients to either block method. Sealed envelopes will be provided to the anesthesiologists, who will apply the block indicated in the envelope at the end of surgery. Both blocks will be performed by experienced anesthesiologists, and only patients operated on under spinal anesthesia will be included in the study.

PENG Block Procedure:

With the patient in the supine position, the ultrasound probe is placed transversely over the anterior superior iliac spine (ASIS). After identifying the ASIS, the transducer is aligned with the pubic ramus and rotated approximately 45 degrees to become parallel to the inguinal crease. The transducer is moved medially until the anterior inferior iliac spine (AIIS), iliopubic eminence (IPE), and psoas tendon are clearly visualized as anatomical landmarks. After confirming the correct location with saline injection, 50 mg of 0.25% bupivacaine will be administered.

QIP Block Procedure:

With the patient in the prone position, a low-frequency convex transducer (2-6 MHz) and a 22G x 100 mm peripheral nerve block needle (Stimuplex® Ultra 360®, B-Braun) will be used. The transducer will be placed transversely at the L3 level to identify the spinal processes, followed by lateral movement to visualize the transverse process within the erector spinae muscle. The transducer will then be rotated parasagittally and moved caudally to locate where the Quadratus Lumborum muscle (QLM) attaches to the iliac crest. After confirming the location with saline, 50 mg of 0.25% bupivacaine will be administered under the fascia of the QLM.

Postoperative Analgesia:

Patients will receive intravenous patient-controlled analgesia (PCA) with 2 mg/mL Tramadol HCl in 100 mL NaCl solution, delivered via bolus doses of 20 mg with a 20-minute lockout period and a total dose limit of 200 mg over 4 hours. Pain scores using the visual analog scale (VAS) will be recorded at rest and with movement at 0, 6, 12, and 24 hours. The total opioid consumption and the need for rescue analgesia (50 mg deksketoprofen in 100 mL mediflex over 20 minutes) will also be assessed. Routine administration of 1 g of intravenous paracetamol will be given at 6 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients and their relatives have provided informed consent,
* Patients aged 18 years or older undergoing femoral fracture surgery,
* ASA score of I-III,
* No history of bleeding diathesis,
* No history of anticoagulant use that contraindicates block application according to guidelines,
* No history of neuropathic diseases such as Diabetes Mellitus,
* No known allergy to local anesthetics.

Exclusion Criteria:

* Lack of informed consent from the patient or their relatives,
* Development of complications during the surgical procedure,
* Need for revision surgery,
* Patient's desire to withdraw from the study,
* Patients under the age of 18,
* ASA score of IV or higher,
* Patients with a history of bleeding diathesis,
* History of anticoagulant use that contraindicates block application according to guidelines,
* Emergency surgeries,
* History of allergy to local anesthetics,
* History of neuropathic diseases,
* Inability to comply with patient-controlled analgesia (PCA) systems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
opioid consumption | 1 day
  Opioid consumption in 24 hours will compared between these two block

SECONDARY OUTCOMES:
Visual Analogue Scale | 1 day
  Visual Analogue Scale scores (0-10) of tge patients will be compared between these two groups in 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No